CLINICAL TRIAL: NCT01627106
Title: A Multicentered, Randomized, Open-Label, Pragmatic Use Study Comparing Vernakalant Therapy to Amiodarone Therapy in Acute Management of Recent Onset Atrial Fibrillation
Brief Title: A Study Comparing Vernakalant Therapy to Amiodarone Therapy in Acute Management of Recent Onset Atrial Fibrillation (AF) (MK-6621-055)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6621-055
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vernakalant (Experimental)
  Interventions: Drug: Vernakalant
- Amiodarone (Active Comparator)
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Vernakalant — Initial intravenous (IV) dose of 3 mg/kg (up to a maximum of 339 mg) over 10 minutes, followed by a 15 minute observation period and, if conversion to sinus rhythm does not occur within 15 minutes of the initial infusion, a second 10 minute infusion of vernakalant at a dose of 2 mg/kg (up to a maximum of 226 mg) will be administered.
  Other Names: Brinavess
  Arms: Vernakalant
Drug: Amiodarone — Administered IV as per product label
  Other Names: Pacerone; Cordarone
  Arms: Amiodarone

SUMMARY:
This study will compare vernakalant therapy to amiodarone therapy in the acute management of recent onset atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic AF (duration of current episode is ≤7 days), which is hemodynamically stable, and participant has no other condition at the time of screening that may result in acute hospitalization
* If female and of reproductive potential, the patient agrees to remain abstinent or use 2 acceptable methods of birth control from time of screening until 30-day follow-up.
* Weigh at least 45 kg
* Receiving adequate anticoagulant therapy

Exclusion Criteria:

* Hypersensitivity to the vernakalant or amiodarone or to citric acid, sodium chloride, sodium hydroxide, or iodine
* Severe aortic stenosis
* Systolic blood pressure <100 mmHg
* New York Heart Association (NYHA) Class III or IV heart failure
* Severe bradycardia, sinus node dysfunction, or second and third degree heart block in the absence of a pacemaker
* Use of IV rhythm control anti-arrhythmics (Class I and III) within 4 hours of study drug administration
* Acute coronary syndrome (including myocardial infarction) within previous 30 days
* History of thyroid dysfunction
* Severe acute respiratory failure or cardiovascular collapse
* Participating in another drug study or has received an investigational drug within 30 days prior to enrollment
* Pregnant or breast-feeding, or expecting to conceive from time of screening until 30-day follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants discharged from the emergency room (ER) to home, home-equivalent, or long-term care facility (LTCF) within 12 hours from randomization | Up to 12 hours from randomization

SECONDARY OUTCOMES:
Number of participants admitted to hospital directly from the ER after randomization | Day 1 (time of ramdomization)